CLINICAL TRIAL: NCT06242184
Title: Post-operative Sensitivity in Composites Using Bacillus Subtilis Procured Novel Nano-fortified Adhesive: a Triple-blind Study
Brief Title: Post-operative Sensitivity in Resin Composites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, NEHAL AMIR, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAMIR
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Caries,Dental; Sensitivity, Tooth
MeSH Terms: conditions — Dental Caries; Dentin Sensitivity | interventions — Nanoparticles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Nano-fortified Adhesive) (Experimental): Titanium dioxide nanoparticles incorporated in dentin adhesive
  Interventions: Procedure: Group A(Nano-fortified Adhesive)
- Group B (Adhesive without Nanoparticles) (Experimental): Adhesive without nanoparticles
  Interventions: Procedure: Group B(Adhesive without nanoparticles)

INTERVENTIONS:
Procedure: Group A(Nano-fortified Adhesive) — Nano-fortified dentin adhesive
  Arms: Group A (Nano-fortified Adhesive)
Procedure: Group B(Adhesive without nanoparticles) — Conventional adhesives without nanoparticles
  Arms: Group B (Adhesive without Nanoparticles)

SUMMARY:
This triple-blind, randomized clinical trial was conducted at the department of Operative dentistry. A total of 60 participants were recruited and were randomly distributed into two groups A and B. After informed consent, restorative treatment was performed. In group A, adhesive with nanoparticles was used for composite restoration while in group B, adhesive without nanoparticles was utilized. Post-operative sensitivity was recorded using VAS score.

DETAILED DESCRIPTION:
Triple-blind, randomized trial, parallel group with an allocation ratio 1:1. A total of 60 participants were recruited from the outpatient department and were randomly distributed into two groups (n=30). After informed consent, restorative treatment was accomplished using an etch and rinse adhesive strategy. In group A , titanium dioxide nano-fortified adhesive was used while in group B, adhesive without nanoparticles was utilized for composite restoration. Post-operative sensitivity was evaluated at follow-up period: one day, one week, two weeks and one month. Visual Analogue scale score was used to record the sensitivity status at follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* participants with goof general health status
* Class I and II primary Carious lesion with a minimum cavity depth of 3 to 5 mm.
* Vital and Periodontally sound teeth

Exclusion Criteria:

* Patient with Temporomandibular dysfunction
* History of spontaneous pain
* Endodontically treated teeth
* Patient on analgesics within the past two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Post-operative sensitivity | One month
  Post-operative sensitivity evaluated at follow-up periods: one day, one week, two weeks and one month using Visual Analogue Scale score with the score 0( none) and score 3( severe sensitivity)

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Amir, BDS, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad
Locations (1):
- School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboelenein AZ, Riad MI, Haridy MF. Effect of a Self-Etch Adhesive Containing Nanobioglass on Postoperative Sensitivity of Posterior Composite Restorations - A Randomized Trial. Open Access Maced J Med Sci. 2019 Jul 25;7(14):2313-2320. doi: 10.3889/oamjms.2019.585. eCollection 2019 Jul 30. PMID 31592280
- [Derived] Amir N, Mansoor A, Eeman N, Ahmed MN, Mansoor E, Hussain K, Palma PJ. Postoperative sensitivity of composites using novel Bacillus subtilis nanofortified adhesives: a triple-blind study. BMC Oral Health. 2024 Sep 12;24(1):1077. doi: 10.1186/s12903-024-04825-2. PMID 39267015